CLINICAL TRIAL: NCT05799196
Title: The Effectiveness of the Microfracture Technique in the Meniscal Healing Rate in Patients With Meniscal Tear Among Indonesian Population
Brief Title: The Effectiveness of the Microfracture Technique in the Meniscal Healing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Leonard Christianto Singjie, Principal Investigator, Hasanuddin University
Other Study IDs: HasanuddinU/Ortopedi/001
Record Dates: First submitted 2023-03-09; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Microfractures; Meniscus Tear
Keywords: meniscus tear; microfracture
MeSH Terms: conditions — Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Microfracture: The patient with meniscus tear would be performed meniscus repair with additional microfracture
  Interventions: Procedure: Microfracture
- Conventional: The patient with meniscus tear would be performed meniscus repair
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Procedure: Microfracture — Microfracture was made in the non-weight bearing chondral to provide the release of MSC and growth factor.

SUMMARY:
Meniscus injuries are a very common cause of knee pain. The meniscus is a semilunar fibrocartilage structure found on the medial and lateral sides of the knee. The meniscus serves to absorb impact and protect the articular cartilage during weight-bearing activities, joint stability, proprioception, and nutrition. This has a significant effect on knee biomechanics.

After the menisci are injured, the biomechanics of the knee change so that degenerative changes occur more frequently in the tibiofemoral compartment. Improvement of tibiofemoral arthrosis after meniscectomy surgery has been demonstrated in several long-term clinical studies. With increasing awareness of the importance of the meniscus in knee biomechanics, various meniscus repair techniques have been developed. In addition, several adjuvants for healing have been proposed to enhance meniscus healing. However, a study showed the meniscal repair failure rate increased from 22% to 24% at 5 years.

Study found the healing rate of meniscus repair, which was accompanied by ACL repair, had a greater healing rate, 93% vs. 50%. Hemarthrosis that occurs after bony tunneling during ACL reconstruction provides a fibrin clot and an environment rich in factors that promote healing of the newly repaired meniscus. The fibrin clot provides the structural foundation for meniscus healing. Transmission factors, such as fibronectin and growth factors, are also present.

Microfracture is a common procedure used for the treatment of damage to the articular cartilage in the knee. This procedure is used to stimulate the production of fibrocartilage in areas of injured cartilage. Microfractures are performed by creating 1 or more small channels (1 to 3 mm in size) that pierce the subchondral bone and release bone-forming components into the joint. Microfractures serve to promote the formation of fibrocartilage over damaged cartilage. Research in 2016 used an animal model (Capra hircus) to investigate the effectiveness of the microfracture technique on meniscus tear healing rates. They found significant healing in meniscal repair accompanied by microfracture technique (65% vs 12%).

However there is still not enough research regarding the efficacy of microfracture in meniscal healing, especially among Indonesian. Therefore, the investigators aim to investigate its efficacy.

ELIGIBILITY:
Inclusion Criteria

1. Patients with meniscus tears
2. The patient underwent meniscus repair surgery using arthroscopy.
3. Have an MRI examination before and after surgery within 6 months post-surgery.

B. Exclusion Criteria

1. Patients with meniscus tears in the white-white area
2. The patient underwent meniscus repair surgery without using arthroscopy
3. The patient did not perform an MRI examination before after surgery within 6 months post-surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with meniscus tear in Wahidin Sudirohusodo General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Healing Rate | 3 months
  Healing Rate, Investigated by MRI and Arthroscopy
Healing Rate | 6 months
  Healing Rate, Investigated by MRI and Arthroscopy

SECONDARY OUTCOMES:
Functional Outcome | 3 months
  Functional Outcome assessed with IKDC ScoreFunctional Outcome assessed with IKDC Score. The higher the score, the higher the level of function and the lower the level of symptoms. A score of 100 suggests no limitation with activities of daily living or sports activities and the absence of symptoms.
Functional Outcome | 6 months
  Functional Outcome assessed with IKDC Score. The higher the score, the higher the level of function and the lower the level of symptoms. A score of 100 suggests no limitation with activities of daily living or sports activities and the absence of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Sakti, MD, Ph.D, Study Chair — Hasanuddin University
Locations (1):
- Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided